CLINICAL TRIAL: NCT00482144
Title: Comparison of the Effectiveness of the Pulsed Dye Laser 585nm Versus 595nm in the Treatment of New Surgical Scars
Brief Title: Study of the Effects of the Pulsed-dye Laser at 585nm and 595nm to Treat Post-operative Scars on Suture-removal Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1999-0694
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Cicatrix; Scars
Keywords: Pulsed-Dye Laser
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment: PDL 450 microseconds (Active Comparator): The scar will be randomly divided into three equal fields. One third of the scar will receive PDL using a 7 mm spot size at 4.0 J (Joules) for 450 microseconds. First treatment will be immediately after suture removal, and then monthly for 3 months.
  Interventions: Procedure: PDL 450 microseconds
- Treatment: PDL 1.5 milliseconds (Active Comparator): The scar will be randomly divided into three equal fields. One third of the scar will receive PDL using a 7 mm spot size at 4.0 J (Joules) for 1.5 milliseconds. First treatment will be immediately after suture removal, and then monthly for 3 months.
  Interventions: Procedure: PDL 1.5 milliseconds
- Control (No Intervention): The scar will be randomly divided into three equal fields. One third of the scar will not receive treatment

INTERVENTIONS:
Procedure: PDL 450 microseconds — The scar will be randomly divided into three equal fields. One third of the scar will receive PDL 585 nm using a 7 mm spot size at 4.0 J (Joules) for 450 microseconds. First treatment will be immediately after suture removal, and then monthly for 3 months.
  Arms: Treatment: PDL 450 microseconds
Procedure: PDL 1.5 milliseconds — The scar will be randomly divided into three equal fields. One third of the scar will receive PDL 585 nm using a 7 mm spot size at 4.0 J (Joules) for 1.5 milliseconds. First treatment will be immediately after suture removal, and then monthly for 3 months.
  Arms: Treatment: PDL 1.5 milliseconds

SUMMARY:
The purpose of this study is to compare the effects of the pulsed-dye laser (PDL) at two different wavelengths, 585nm and 595nm, in the treatment of post-surgical scars starting on suture-removal day.

DETAILED DESCRIPTION:
Many treatment modalities have been used for the treatment of scars such as dermabrasion, cryotherapy, intralesional corticosteroids, surgical scar revision, and lasers, among others. Previous studies have shown that treatment of scars with the pulsed dye laser (PDL) alone or in combination with other modalities (e.g. corticosteroids, 5-Fluoruracil, silicone sheets) improves the vascularity, pliability, color, and height of hypertrophic scars and keloids. Currently, the PDL has become the laser of choice for the treatment of scars.

To our knowledge, there are no reports in the literature comparing the effects of different wavelengths of the PDL for the treatment of scars. The objective of this study was to compare the effects of the PDL at 585nm vs 595nm in the treatment of postsurgical linear scars starting the day of suture removal.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Postoperative linear scars greater than 6 cm
* Skin photo-types I-IV

Exclusion Criteria:

* Patient should not be taking any systemic, topical, or intralesional treatment of the scars

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-07; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale Visual Analog Scale | 9 months

SECONDARY OUTCOMES:
Visual Analog Scale | 9 months
Blinded Evaluator assessments | 9 months
  The scar section will be compared in terms of: Pigmentation 0 normal color, close to normal skin 1 hypopigmentation 2 hyperpigmentation Vascularity 0 normal color, close to normal skin 1 pink, slight increase in blood supply 2 red, significant increase in blood supply 3 purple, excessive increase in blood supply Pliability 0 normal, normal pliability 1 supple, flexible with minimal resistance 2 yielding, giving way to pressure 3 firm, solid, inflexible unit 4 banding, rope-like tissue that blanches with extension of scar 5 contracture, permanent shortening Height 0 normal, flat 1 <2 mm 2 <5 mm 3 >5 mm

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida, United States

REFERENCES:
- [Background] Nouri K, Jimenez GP, Harrison-Balestra C, Elgart GW. 585-nm pulsed dye laser in the treatment of surgical scars starting on the suture removal day. Dermatol Surg. 2003 Jan;29(1):65-73; discussion 73. doi: 10.1046/j.1524-4725.2003.29014.x. PMID 12534515